CLINICAL TRIAL: NCT00771953
Title: 0822GCC Randomized, Double-Blind, Placebo-Controlled Multicenter Phase 2 Study of the Efficacy and Safety of Apricoxib in Combination With Either Docetaxel or Pemetrexed in Non-Small Cell Lung Cancer Patients
Brief Title: 0822GCC: Phase 2 Study of Efficacy and Safety of Apricoxib/Placebo With Docetaxel or Pemetrexed in Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Tragara Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HP-00043076; 0822GCC; UMGCC 0822 (Other: University of Maryland Greenebaum Cancer Center)
Record Dates: First submitted 2008-10-10; First posted 2008-10-15 (Estimated); Results first posted 2013-07-22 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Lung Cancer; Non Small Cell Lung Cancer
Keywords: apricoxib; docetaxel; pemetrexed; Stage IIIb or Stage IV
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — apricoxib; Docetaxel; Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apricoxib (Experimental): Apricoxib 400mg once a day
  Interventions: Drug: apricoxib; Drug: Docetaxel or Pemetrexed
- Placebo (Placebo Comparator): Placebo once a day
  Interventions: Drug: Placebo; Drug: Docetaxel or Pemetrexed

INTERVENTIONS:
Drug: apricoxib — Oral apricoxib tablets will be provided as white or off-white film-coated tablets available in 100mg strength to be taken every day
  Arms: Apricoxib
Drug: Placebo — Oral placebo tablets will be provided as white or off-white film-coated tablets to be taken every day
  Arms: Placebo
Drug: Docetaxel or Pemetrexed — Docetaxel 75mg/m2 or Pemetrexed 500mg/m2 given as an IV infusion every 21 days. TheTreating physician will determine chemotherapy drug as per his usual practice.

SUMMARY:
The primary objective is to determine the anti-tumor activity of the combination of apricoxib + either docetaxel (AP/DC) or pemetrexed (AP/PE) compared with placebo + either docetaxel (P/DC) or pemetrexed (P/PE) as measured by progression free survival in patients with Stage IIIb (pleural effusion)or Stage IV non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
Patients diagnosed with advanced non-small cell lung cancer that has not responded to platinum-based chemotherapy are eligible to particvpate in this study.

Current standard treatments for this type of lung cancer are generally not effective in preventing the cancer from growing. The purpose of this study is to see if adding the drug apricoxib to standard chemotherapy is effective in treting NSCLC. Apricoxib is an investigational drug. Investigational means that it is not approved by the Food and Drug Administration (FDA). Laboratory studies suggest that apricoxib may be useful in the treatment of cancer . This is seen particularly when it is combined with chemotherapy drugs. However, this has not been proven in humans.

Laboratory evidence indicates that apricoxib may benefit patients whose disease over-produces a substance called COX-2. COX-2 can be detected in the urine as a substance called PGE-M (prostaglandin E metabolite). It is thought that patients who have a PGE-M level in the urine that decreases by at least half after taking apricoxib may benefit more than patients whose urine PGE-M decreases by less than half after apricoxib.

This study evaluated whether adding apricoxib to standard chemotherapy treatment will improve outcomes in patients with non-small cell lung cancer whose urine PGE-M decreases at least 50% after taking apricoxib. Apricoxib or placebo was added to either docetaxel or pemetrexed treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically determined stage IV non-small cell lung cancer (NSCLC), including stage IIIb (pleural effusion) (histology or cytology acceptable).
* Documented progression after 1 prior platinum-based chemotherapy. No more than one prior chemotherapy regimen is permitted. Patients may have also received erlotinib (before, after or concurrently with platinum based therapy).
* Measurable disease by RECIST criteria
* Age at least 18 years.
* ECOG performance status of 0-2.
* Required Laboratory Values (within 28 days before randomization) :

  * Hb ≥ 9.0gm/dL; transfusions permitted
  * ANC ≥ 1500/mm3
  * Platelets ≥ 100,000/mm3
  * INR ≤ 1.5
  * Serum creatinine (Cr) within normal limits for laboratory OR Creatinine clearance greater than or equal to 45 ml/min. 24 hour measured CCr is also acceptable (calculated by the Cockcroft and Gault equation).
  * SGOT and SGPT < 2 X the ULN; if liver metastases are present then must be < 5 X the ULN
  * Bilirubin ≤ Institutional ULN
  * Albumin ≥ or equal to 2.5 mg/dl
* May have been treated with anti-EGFR kinase therapy in addition to a platinum based therapy or concurrently with platinum therapy.
* Provide written informed consent and HIPAA authorization and agree to abide by the study restrictions and return for the required assessments.
* Women of child-bearing potential must have negative pregnancy test (serum B-HCG) with a sensitivity of at least 50 mIU/L within 7 days prior to the initiation of treatment and must have used effective contraception (recommended to be two reliable forms of contraception used simultaneously) or must have been sexually abstinent for at least 4 weeks prior to the negative pregnancy test through entry in the study.
* Female patients and male patients with female partners of child-bearing potential must agree to sexual abstinence or to practice effective contraception (recommended to be two reliable forms of contraception used simultaneously). At least one non-hormonal method strongly recommended. Male patients with female sexual partners who are pregnant, or of childbearing potential must agree to use condoms during and for at least 1 month after the last dose of apricoxib.

Exclusion Criteria:

* Pregnant or breast feeding
* Known hypersensitivity to apricoxib, docetaxel, other drugs formulated with polysorbate 80, pemetrexed, sulfonamides, aspirin, or other NSAIDs.
* Radiation therapy within 2 weeks or chemotherapy within 3 weeks or non-cytotoxic investigational agents within 3 weeks of initiating study treatment or patients who have not recovered from adverse effects due to agents administered > 3 weeks prior to initiating study treatment. Screening for urinary PGE-M suppression may begin during this time period.
* Evidence of New York Heart Association class III or greater cardiac disease. History of myocardial infarction, stroke, ventricular arrhythmia, or symptomatic conduction abnormality within 12 months.
* Concurrent severe or uncontrolled medical disease that could compromise the safety of the patient or compromise the ability of the patient to complete the study.
* Known HIV infection or AIDS. Testing not required.
* Symptomatic central nervous system metastases; the patient must be stable after radiotherapy for ≥ 2 weeks. Patients must be off all steroid or antiseizure medications for this indication for ≥ 2 weeks. Patients with CNS metastases that are untreated are eligible if there is no evidence of midline shift, requirement for steroids or antiseizure medications or neurologic symptoms.
* History of upper GI bleeding, ulceration, or perforation within the past 5 years.
* Concurrent use of COX-2 inhibitors or other NSAIDs for 2 days prior to the first dose of study treatment and during study, including aspirin for 7 days prior to the first dose of study treatment and during study.
* Previous COX-2 inhibitor therapy for this diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2008-11; Primary Completion 2012-05 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin J Edelman, Principal Investigator — University of Maryland Greenebaum Cancer Center
Locations (12):
- United States (12):
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Mercy Research Institute, Miami, Florida
  - University of Miami, Miami, Florida
  - Rush University Medical Center, Chicago, Illinois
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Weill Medical Cornell University, New York, New York
  - Stony Brook Cancer Center (SUNY), Stony Brook, New York
  - Providence Portland Medical Center, Portland, Oregon
  - Abramson Cancer Center of Uof Pennsylvania, Philadelphia, Pennsylvania
  - West Virginia University Clinical Trials Research Unit, Morgantown, West Virginia

REFERENCES:
- [Background] Rao PN, Grover RK. Apricoxib, a COX-2 inhibitor for the potential treatment of pain and cancer. IDrugs. 2009 Nov;12(11):711-22. PMID 19844858
- [Background] Edelman MJ, Watson D, Wang X, Morrison C, Kratzke RA, Jewell S, Hodgson L, Mauer AM, Gajra A, Masters GA, Bedor M, Vokes EE, Green MJ. Eicosanoid modulation in advanced lung cancer: cyclooxygenase-2 expression is a positive predictive factor for celecoxib + chemotherapy--Cancer and Leukemia Group B Trial 30203. J Clin Oncol. 2008 Feb 20;26(6):848-55. doi: 10.1200/JCO.2007.13.8081. PMID 18281656
- [Background] Reckamp KL, Krysan K, Morrow JD, Milne GL, Newman RA, Tucker C, Elashoff RM, Dubinett SM, Figlin RA. A phase I trial to determine the optimal biological dose of celecoxib when combined with erlotinib in advanced non-small cell lung cancer. Clin Cancer Res. 2006 Jun 1;12(11 Pt 1):3381-8. doi: 10.1158/1078-0432.CCR-06-0112. PMID 16740761
- [Background] Murphey LJ, Williams MK, Sanchez SC, Byrne LM, Csiki I, Oates JA, Johnson DH, Morrow JD. Quantification of the major urinary metabolite of PGE2 by a liquid chromatographic/mass spectrometric assay: determination of cyclooxygenase-specific PGE2 synthesis in healthy humans and those with lung cancer. Anal Biochem. 2004 Nov 15;334(2):266-75. doi: 10.1016/j.ab.2004.08.019. PMID 15494133
- [Background] Gitlitz BJ, et al. Apricot-l: Results of a biomarker-based phase II randomized placebocontrolled study of apricoxib in combination with erlotinib in non-small cell lung cancer (NSCLC) patients. Journal of Clinical Oncology 29: 2011 (suppl; abstr 7528)
- [Background] Groen HJ, Sietsma H, Vincent A, Hochstenbag MM, van Putten JW, van den Berg A, Dalesio O, Biesma B, Smit HJ, Termeer A, Hiltermann TJ, van den Borne BE, Schramel FM. Randomized, placebo-controlled phase III study of docetaxel plus carboplatin with celecoxib and cyclooxygenase-2 expression as a biomarker for patients with advanced non-small-cell lung cancer: the NVALT-4 study. J Clin Oncol. 2011 Nov 10;29(32):4320-6. doi: 10.1200/JCO.2011.35.5214. Epub 2011 Oct 11. PMID 21990410
- [Background] Markowitz SD. Aspirin and colon cancer--targeting prevention? N Engl J Med. 2007 May 24;356(21):2195-8. doi: 10.1056/NEJMe078044. No abstract available. PMID 17522404
- [Derived] Edelman MJ, Tan MT, Fidler MJ, Sanborn RE, Otterson G, Sequist LV, Evans TL, Schneider BJ, Keresztes R, Rogers JS, de Mayolo JA, Feliciano J, Yang Y, Medeiros M, Zaknoen SL. Randomized, double-blind, placebo-controlled, multicenter phase II study of the efficacy and safety of apricoxib in combination with either docetaxel or pemetrexed in patients with biomarker-selected non-small-cell lung cancer. J Clin Oncol. 2015 Jan 10;33(2):189-94. doi: 10.1200/JCO.2014.55.5789. Epub 2014 Dec 1. PMID 25452446

RESULTS

PARTICIPANT FLOW:
Recruitment Details: University Medical Centers and Hospital Based Oncology Programs recruited participants from November 2011 through August 2011
Pre-assignment Details: 110 patients started a 5 day run in period with 400mg apricoxib. 7 did not complete due to AEs, and 23 did not have at least 50% drop in PGE-M (randomization requirement). Of the remaining 80, 2 withdrew, 2 were ineligible by physician discretion, 1 died and 3 had progressive disease. Thus, 72 patients were randomized.
Groups:
- Apricoxib Plus Docetaxel or Pemetrexed: Apricoxib 400mg qd and either docetaxel 75mg/m2 or pemetrexed 500mg/m2 q21 days
- Placebo Plus Docetaxel or Pemetrexed: Placebo and either docetaxel 75mg/m2 or pemetrexed 500mg/m2 q21 days
Period: Overall Study
Arm/Group | Apricoxib Plus Docetaxel or Pemetrexed | Placebo Plus Docetaxel or Pemetrexed
Started | 36 | 36
Completed | 26 | 26
Not Completed | 10 | 10
Not completed — Adverse Event | 5 | 3
Not completed — Death | 2 | 2
Not completed — Progression before active Tx | 1 | 2
Not completed — Sponsor decision | 1 | 0
Not completed — Other complicating disease | 1 | 0
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Apricoxib Plus Docetaxel or Pemetrexed | Placebo Plus Docetaxel or Pemetrexed | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Customized [Median (Full Range); unit: years] | 62 [42 to 87] | 66 [49 to 76] | 64 [42 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: For determining progression-free survival, progression was determined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0). Progression was defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From the date of randomization until the first date that recurrent or progressive disease is objectively documented.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Apricoxib Plus Docetaxel: Apricoxib 400mg qd plus docetaxel 75mg/m2 q21 days
- Placebo Plus Docetaxel: Placebo plus docetaxel 75mg/m2 q21 days
- Apricoxib Plus Pemetrexed: Apricoxib 400mg qd plus pemetrexed 500mg/m2 q21 days
- Placebo Plus Pemetrexed: Placebo plus pemetrexed 500mg/m2 q21 days
Arm/Group | Apricoxib Plus Docetaxel | Placebo Plus Docetaxel | Apricoxib Plus Pemetrexed | Placebo Plus Pemetrexed
Number analyzed (Participants) | 17 | 20 | 19 | 16
days | 75 [47 to 104] | 97 [48 to 216] | 103 [62 to 225] | 98 [37 to 197]

ADVERSE EVENTS:
Arm/Group | Apricoxib Plus Docetaxel or Pemetrexed | Placebo Plus Docetaxel or Pemetrexed
Serious Adverse Events (participants affected / at risk) | 11/36 | 11/36
Other Adverse Events (participants affected / at risk) | 12/36 | 11/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apricoxib Plus Docetaxel or Pemetrexed (N=36) | Placebo Plus Docetaxel or Pemetrexed (N=36)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — progressive disease
Abdominal pain (General disorders) | 0 (0) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
Aseptic meningitis (Nervous system disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
CPOD exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Coumadin toxicity (General disorders) | 1 (1) | 0 (0)
Creatinine increase (Hepatobiliary disorders) | 0 (0) | 1 (1)
Dehydration (General disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Granulocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 1 (1) | 1 (1)
Hyperkalemia (General disorders) | 1 (2) | 0 (0)
Hypernatremia (General disorders) | 0 (0) | 1 (1)
Hypoglycemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyponatremia (General disorders) | 0 (0) | 1 (1)
Hypoxia (General disorders) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Thrombosis (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apricoxib Plus Docetaxel or Pemetrexed (N=36) | Placebo Plus Docetaxel or Pemetrexed (N=36)
Hyponatremia (General disorders) | 2 (3) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 9 (9) | 9 (10)
Lowered WBC count (Blood and lymphatic system disorders) | 2 (3) | 1 (1)

LIMITATIONS AND CAVEATS:
This study is limited by the relatively low numbers and the hetereogeneity between concurrent treatments (docetaxel vs. pemetrexed). However, in analyses stratified by docetaxel and pemetrexed, results for an affect of apricoxib were still null.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes